CLINICAL TRIAL: NCT01655693
Title: Multicentre, Randomised, Controlled, Open-label Study Comparing the Efficacy and Safety of Doxorubicin Transdrug™ to Best Standard of Care in Patients With Advanced Hepatocellular Carcinoma. ReLive Study.
Brief Title: Efficacy and Safety Doxorubicin Transdrug Study in Patients Suffering From Advanced Hepatocellular Carcinoma
Acronym: ReLive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA2011/03/04; 2011-002843-92 (EudraCT Number)
Record Dates: First submitted 2012-07-26; First posted 2012-08-02 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Intermediate/advanced hepatocellular carcinoma; After failure or intolerance to Sorafenib.
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Doxorubicin Transdrug (DT) at 20 mg/m2 (Experimental): DT will be infused over 6 hours through the intravenous (IV) route at dose of 20 mg/m2 on Day 1 and will be repeated every 4 weeks until disease progression or unacceptable toxicity
  Interventions: Drug: Doxorubicin 20 mg/m2
- Doxorubicin Transdrug (DT) at 30 mg/m2 (Experimental): DT will be infused over 6 hours through the IV route at dose of 30 mg/m2 on Day 1 and will be repeated every 4 weeks until disease progression or unacceptable toxicity
  Interventions: Drug: Doxorubicin 30 mg/m2
- Best Standard of Care (Active Comparator): Patients randomized in the control group will receive treatment according to the investigator's choice, until disease progression or unacceptable toxicity
  Interventions: Drug: Best Standard of Care

INTERVENTIONS:
Drug: Doxorubicin 20 mg/m2
  Other Names: Doxorubicin Transdrug (DT) at 20 mg/m2
  Arms: Doxorubicin Transdrug (DT) at 20 mg/m2
Drug: Doxorubicin 30 mg/m2
  Other Names: Doxorubicin Transdrug (DT) at 30 mg/m2
  Arms: Doxorubicin Transdrug (DT) at 30 mg/m2
Drug: Best Standard of Care
  Other Names: BSC
  Arms: Best Standard of Care

SUMMARY:
The purpose of this phase III study is to determine whether Doxorubicin Transdrug (DT) is effective in the treatment of patients suffering from advanced Hepatocellular Carcinoma (HCC) after failure or intolerance to Sorafenib. Patients with HCC with or without cirrhosis and with good liver functions are eligible. Only those who can not benefit from treatment for which efficacy is demonstrated are eligible.

These patients are usually proposed either best standard of care (BSC) or participation to clinical trials. Patients eligible for the RELIVE study will receive either DT at 20 mg/m2 or DT at 30 mg/m2 or the BSC.

DETAILED DESCRIPTION:
Doxorubicin-Transdrug™ (DT) is a nanoparticle formulation of doxorubicin.In in vitro and in vivo models, DT was shown to overcome the multidrug resistance (MDR) and to be more effective than doxorubicin on both sensitive and resistant tumour models and in particular in the X/myc bi-transgenic MDR murine model of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breast feeding female;
* Aged ≥ 18 years;
* Patient with:

  * advanced HCC (BCLC-C according to BCLC staging classification) having progressed under Sorafenib therapy or intolerant to Sorafenib, or;
  * intermediate HCC (BCLC-B) non eligible or non responders to transarterial chemoembolization (TACE), and having progressed under or intolerant to Sorafenib therapy
* Patients with porta hepatis lymph nodes, extrahepatic metastases, or portal/suprahepatic vein thrombosis without extension in inferior/superior vena cava, are eligible;
* HCC diagnosed according to the American Association for Study of Liver Diseases (AASLD) and/or European Association for the Study of the Liver (EASL) criteria:

  * Radiological Criteria applicable in cirrhotic liver:
* Nodule ≥ 10 mm: one imaging technique among MRI and CT-scan showing typical appearances for HCC defined as arterial enhancement and rapid washout in portal venous or delayed phase;
* If appearance not typical for HCC on initial imaging: second contrast enhanced study (CT or MRI) showing typical appearances for HCC defined as arterial enhancement and rapid wash-out in portal venous or delayed phase;

  * And/Or cyto-histology criteria (e.g. in case of atypical lesions for HCC at imaging, absence of cirrhosis);
* Without cirrhosis or with a non decompensated cirrhosis (Child-Pugh score from A5 to B7 included);
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1;
* Laboratory tests as follows:

  * Platelets ≥ 50,000 /mm3
  * Neutrophil count ≥ 1000/mm3
  * Hemoglobin ≥ 10g/dL
  * Serum transaminases < 5 upper limit normal (ULN) (NCI/common toxicity criteria (CTC) grades 0, 1, or 2)
  * Alkaline phosphatases < 5 ULN (NCI/CTC grades 0, 1, or 2)
  * Serum bilirubin < 35 micromolar (µM)/L (or 2.0 mg/dL);
* Signed and dated written informed consent form.

Exclusion Criteria:

* Cirrhosis with a Child-Pugh score B8-C15;
* Untreated chronic hepatitis B;
* Patients eligible for curative treatments (transplantation, surgical resection, percutaneous treatment);
* Patients eligible for palliative treatments with demonstrated efficacy: TACE, Sorafenib; Patients who failed to Sorafenib treatment or intolerant to sorafenib are eligible and can be included if Sorafenib has been stopped at least 2 weeks before randomization;
* Prior history of malignancy with the exception of adequately treated basal cell carcinoma or in situ cervical cancer in complete remission since five years at least;
* HCC developed on transplanted liver;
* HIV infection;
* Risk of variceal bleeding;
* Oxygen saturation (SaO2) < 95%;
* Presence of a significant acute or chronic respiratory disease defined as NCI/CTCAE > grade 2;
* Presence of recent (< 6 months) or current cardiac failure (class III or IV New York Heart Association (NYHA) classification), recent (< 6 months) acute coronary syndrome, clinically significant ECG abnormalities or recent (less than 6 months) acute vascular diseases (stroke, myocardial infarction (MI)…);
* Prior cumulative dose of 300 mg/m² of doxorubicin or equivalent;
* Patients currently treated with immunosuppressive agents that cannot be stopped;
* Patients whose medical or surgical conditions are unstable and may not allow the study completion or compliance, and specially patients with uncontrolled diabetes;
* Uncontrolled systemic infection;
* Patients with a life expectancy of less than 2 months;
* Patients who have received an experimental drug in another clinical trial in the last 30 days prior to randomization in the present clinical trial;
* Women of child-bearing age who are unwilling or unable to use an effective contraception method during the study treatment period and for 6 months after the last administration of study drug, and their male partner(s) refusing to use a condom (if applicable);
* Men who are unwilling or unable to use a condom during the study treatment period and for 6 months after the last administration of study drug, and their female partner(s) refusing to use one of the appropriate effective contraception methods (if applicable);
* Patients unwilling or unable to comply with protocol requirements and scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Merle, MD, Principal Investigator — Croix-Rousse Hospital - Lyon-France
Locations (70):
- United States (3):
  - Gabrail Cancer Center, Canton, Ohio
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
- Austria (2):
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Medical University Vienna, Vienna
- Belgium (4):
  - CHU Brugmann, Brussels
  - UCL Saint-Luc, Brussels
  - CHU Sart Tilman, Liège
  - CHU UCL Mont-Godinne Dinant, Yvoir
- Egypt (6):
  - Medical Oncology department /Mansoura University Hospitals, Al Mansurah
  - Clinical Research Center/ Alexandria university hospital, Alexandria
  - Oncology Department, Medical Research Institute, Alexandria University, Alexandria
  - Medical Oncology department /Ain Shams University Hospitals, Cairo
  - National hepatology and tropical medicine research institute, Cairo
  - National Liver Institute / Menoufyia University, Menofia
- France (25):
  - Hospital Amiens, Amiens
  - Hospital Jean Minjoz, Besançon
  - Hospital Saint André, Bordeaux
  - Centre hospitalier P Oudot, Bourgoin
  - Hospital Estaing, Clermont-Ferrand
  - Centre Hospitalier Beaujon, Clichy
  - Hospital Henri-Mondor, Créteil
  - Centre Jean-François Leclerc, Dijon
  - CHU, Dijon
  - Hospital Grenoble, La Tronche
  - CHU Dupuytren, Limoges
  - Hospital Croix Rousse, Lyon
  - Hospital La Timone, Marseille
  - Hospital Saint Eloi, Montpellier
  - Hospital Brabois, Nancy
  - Hospital Hotel Dieu, Nantes
  - CHU - Hôpital Archet, Nice
  - Hospital La Source, Orléans
  - Hospital Pitié-Salpetriere, Paris
  - Hospital Tenon, Paris
  - Hospital Saint Jean, Perpignan
  - CHU de Rouen- Hôpital Charles Nicolle, Rouen
  - IC LOIRE, Saint-Etienne
  - Hospital Civil, Strasbourg
  - Hospital Paul Brousse, Villejuif
- Germany (5):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universität Leipzig AöR, Leipzig
  - Klinikum rechts der Isar der TU Munchen II, München
- Hungary (4):
  - Semmelweis Egyetem Radiológiai és Onkoterápiás Klinika, Budapest
  - Egyesített Szent István és Szent László Kórház - Rendelőintézet, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum Onkológiai Intézet, Debrecen
  - Szegedi Tudományegyetem Onkoterápiás Klinika, Szeged
- Italy (8):
  - Irccs Centro Di Riferimento Oncologico (Cro), Aviano
  - Ospedale Civile e degli Infermi, Faenza
  - Ausl 12 Livorno Ospedale Unico della Versilia, Lido di Camaiore
  - IRST Istituto Romagnolo Ricerca e Cura dei Tumori, Meldola
  - Granda Osp. Magg. Policlinico, Milan
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - A.O. Ospedale Maggiore della Carità, Novara
  - Rimini
- Ain Wazein Hospital, El Chouf, Lebanon
- Spain (10):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Virgen de la Arrixaca, El Palmar Murcia
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital General Universario Gregorio Maranon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Universario Son Espaces, Palma de Mallorca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Río Hortega, Valladolid
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Ege Univeristy Medical Faculty,, Izmir

REFERENCES:
- [Derived] Merle P, Blanc JF, Phelip JM, Pelletier G, Bronowicki JP, Touchefeu Y, Pageaux G, Gerolami R, Habersetzer F, Nguyen-Khac E, Casadei-Gardini A, Borbath I, Tran A, Wege H, Saad AS, Colombo M, Abergel A, Richou C, Waked I, Yee NS, Mole A, Attali P, Le Boulicaut J, Vasseur B; RELIVE Investigators. Doxorubicin-loaded nanoparticles for patients with advanced hepatocellular carcinoma after sorafenib treatment failure (RELIVE): a phase 3 randomised controlled trial. Lancet Gastroenterol Hepatol. 2019 Jun;4(6):454-465. doi: 10.1016/S2468-1253(19)30040-8. Epub 2019 Apr 4. PMID 30954567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 541 patients were screened, and 397 patients were randomized a 1:1:1 allocation at 69 sites in 11 countries worldwide. The randomization was performed using an interactive web response system (IWRS) with stratification based on region.
  Enrollment of first patient was June 15, 2012. Data cutoff was May 28, 2017 (24 months) for initial study and May 10, 2019, for follow-up period (45 months).
Pre-assignment Details: Of the 144 patients who failed screening, the most common reason for screen failure was meeting liver function exclusion criteria.
Groups:
- Doxorubicin Transdrug (DT) at 20 mg/m2: DT was infused over 6 hours through the intravenous (IV) route at dose of 20 mg/m2 on Day 1 and was repeated every 4 weeks until disease progression or unacceptable toxicity.
- Doxorubicin Transdrug at 30 mg/m2: DT was infused over 6 hours through the IV route at dose of 30 mg/m2 on Day 1 and was repeated every 4 weeks until disease progression or unacceptable toxicity.
- Best Standard of Care: Patients randomized in the control group received treatment according to the investigator's choice, until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care
Started | 130 | 133 | 134
Completed | 4 | 7 | 4
Not Completed | 126 | 126 | 130
Not completed — Progression of Disease | 92 | 76 | 58
Not completed — Death | 8 | 9 | 12
Not completed — Serious Adverse Event | 3 | 15 | 11
Not completed — Withdrawal by Subject | 3 | 2 | 20
Not completed — Adverse Event | 3 | 11 | 3
Not completed — Aggravation of Liver Dysfunction | 5 | 4 | 0
Not completed — Non-Compliance | 0 | 0 | 7
Not completed — No Respect of Criteria for Continuing Treatment | 1 | 3 | 0
Not completed — Protocol Violation | 1 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Screening Failure | 1 | 0 | 0
Not completed — Other | 8 | 6 | 15

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population: all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care | Total
Number analyzed (Participants) | 130 | 133 | 134 | 397
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 62 | 57 | 169
  >=65 years | 80 | 71 | 77 | 228
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 27 | 18 | 57
  Male | 118 | 106 | 116 | 340
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 120 | 119 | 125 | 364
  Black | 1 | 3 | 2 | 6
  Asian | 1 | 3 | 2 | 6
  Other | 1 | 3 | 3 | 7
  Hispanic or Latino | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  North African | 6 | 2 | 0 | 8
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Unknown | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 3 | 7
  Europe | 118 | 120 | 119 | 357
  Middle East | 10 | 11 | 12 | 33
Alcohol Consumption [Count of Participants; unit: Participants]
  No Significant Alcohol Consumption | 119 | 127 | 123 | 369
  Active Alcohol Consumption | 11 | 6 | 11 | 28
Child Pugh Class [Count of Participants; unit: Participants] — The Child-Pugh score is determined by scoring five clinical measures of liver disease: encephalopathy, ascites, albumin, total bilirubin, prothrombin time rate. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe. The total score is used to assign the Child-Pugh class as follows:
  Class A: 5-6 points (least severe liver disease) Class B: 7-9 points (moderately severe liver disease) Class C: 10-15 points (most severe liver disease)
  Participants
    Child Pugh A | 114 | 109 | 113 | 336
    Child Pugh B | 15 | 24 | 21 | 60
    Child Pugh C | 1 | 0 | 0 | 1
Previous Hepatocellular Carcinoma (HCC) Treatments [Count of Participants; unit: Participants] — Prior treatment for HCC is collected at baseline as part of the medical history for surgery and the following drugs and therapy: sorafenib, hormone therapy, tyrosine kinase inhibitor, investigational drug, cytotoxic chemotherapy, and other anticancer therapy. Patients may have received treatment in more than one of these categories.
  Participants
    Surgery/Resection | 41 | 49 | 40 | 130
    Loco-regional Treatment | 84 | 84 | 84 | 252
    Radiotherapy | 14 | 14 | 9 | 37
    Sorafenib | 130 | 133 | 134 | 397
    Other Systemic Anticancer Therapy | 68 | 73 | 80 | 221
Medical History Active [Count of Participants; unit: Participants] — Active medical history of patient at time of baseline assessment is collected. Presenting all active medical history that occurred at an incidence of >=10% of the patients in at least one of the treatment groups is presented for all groups. Patients may fall into more than one of these categories.
  Participants
    Hypertension | 73 | 82 | 84 | 239
    Type 2 Diabetes Mellitus | 28 | 15 | 35 | 78
    Diabetes Mellitus | 17 | 26 | 17 | 60
    Hypercholestrolaemia | 12 | 14 | 9 | 35
    Varices Oesophageal | 14 | 24 | 15 | 53
    Chronic Obstructive Pulmonary Disease | 13 | 8 | 9 | 30
    Thrombocytopenia | 7 | 15 | 8 | 30
HCC History-Cirrhosis [Count of Participants; unit: Participants]
  Yes | 93 | 96 | 101 | 290
  No | 36 | 35 | 31 | 102
  Unknown | 1 | 2 | 2 | 5
HCC History - Cyto Histology [Count of Participants; unit: Participants] — Used American Association for the Study of Liver Diseases (AASLD)/European Association for the Study of the Liver (EASL) Criteria
  Participants
    Yes | 80 | 87 | 92 | 259
    No | 50 | 46 | 42 | 138
HCC History - Macroscopic Vascular Invasion [Count of Participants; unit: Participants] — Multiple selection possible for vascular invasion.
  Participants
    Macroscopic Portal Vein or Portal Branch Vascular Invasion - Yes | 48 | 41 | 39 | 128
    Macroscopic Portal Vein or Portal Branch Vascular Invasion - No | 82 | 92 | 95 | 269
    Supra-hepatic Vascular Invasion Vein - Yes | 9 | 8 | 10 | 27
    Supra-hepatic Vascular Invasion Vein - No | 121 | 125 | 124 | 370
    Vascular Invasion (Portal and/or Supra Hepatic) - Yes | 50 | 43 | 45 | 138
    Vascular Invasion (Portal and/or Supra Hepatic) - No | 80 | 90 | 89 | 259
HCC History - Extra Hepatic Spread - Porta Hepatic Lymph Nodes [Count of Participants; unit: Participants]
  Yes | 24 | 19 | 31 | 74
  No | 99 | 104 | 98 | 301
  Unknown | 7 | 10 | 5 | 22
HCC History - Extra Hepatic Spread - Distant Metastases [Count of Participants; unit: Participants]
  Yes | 64 | 68 | 71 | 203
  No | 64 | 61 | 57 | 182
  Unknown | 2 | 4 | 6 | 12
HCC History - Aetiology of Underlying Liver Disease [Count of Participants; unit: Participants] — Percentages are based on the number of patients in the respective group. Patients could have more than one aetiology of underlying liver disease and may be counted in more than one category.
  Participants
    Alcohol | 64 | 60 | 68 | 192
    Hepatitis C Virus | 40 | 40 | 38 | 118
    Nonalcoholic Steatohepatitis | 14 | 21 | 23 | 58
    Unknown | 26 | 14 | 16 | 56
    Hepatitis B Virus | 7 | 16 | 14 | 37
    Other | 4 | 12 | 3 | 19
    Hemochromatosis | 3 | 6 | 4 | 13
    Autoimmune | 0 | 0 | 0 | 0
    Primary Biliary Cirrhosis | 0 | 0 | 0 | 0
HCC History - Nodule in the Liver [Count of Participants; unit: Participants]
  Single Nodule | 15 | 5 | 8 | 28
  Multiple Nodules | 102 | 106 | 111 | 319
  Infiltrate HCC | 8 | 17 | 13 | 38
  Unknown | 5 | 5 | 2 | 12
HCC History - Disease Duration [Mean (Standard Deviation); unit: months] — Disease duration is calculated at study entry in months as the screening visit date - cancer diagnosis date.
  months | 28.1 (24.04) | 30.5 (35.86) | 31.5 (28.38) | 30.1 (29.83)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to the date of death from any cause.
Time Frame: Time from date of randomization to the date of death from any cause with initial assessment up to 24 months and follow-up assessment up to 45 months.
Population: Intent-to-treat (ITT) Population: All randomized patients. The DT at 20 mg/m2 and 30 mg/m2 are combined into DT pooled experimental group for comparison with the BSC group. The primary analysis per protocol is DT pooled versus BSC and not individual DT groups.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Doxorubicin Transdrug (DT) 20 mg/m2 Group: DT was infused over 6 hours through the intravenous route at dose of 20 mg/m2 on Day 1 and was repeated every 4 weeks until disease progression or unacceptable toxicity.
- Doxorubicin Transdrug Pooled: The DT 20 mg/m2 and 30 mg/m2 treatment group were pooled together for OS comparison to Best Standard of Care (BCS) for initial study.
- Best Standard of Care (BSC): Patients randomized in the control group received treatment according to the investigator's choice, until disease progression or unacceptable toxicity in initial study.
Arm/Group | Doxorubicin Transdrug (DT) 20 mg/m2 Group | Doxorubicin Transdrug at 30 mg/m2 | Doxorubicin Transdrug Pooled | Best Standard of Care (BSC)
Number analyzed (Participants) | 130 | 133 | 263 | 134
months
  OS up to 24 Months | 10.1 [7.3 to 11.4] | 8.9 [7.0 to 10.3] | 9.1 [8.1 to 10.4] | 9.0 [7.1 to 11.8]
  OS up to 45 Months | 9.8 [7.4 to 11.2] | 8.8 [7.1 to 10.3] | 8.9 [8.1 to 10.3] | 9.0 [7.2 to 11.8]
Statistical Analysis 1: Comparison: Doxorubicin Transdrug (DT) 20 mg/m2 Group vs Doxorubicin Transdrug at 30 mg/m2 vs Doxorubicin Transdrug Pooled vs Best Standard of Care (BSC); Initial 24 month assessment: the primary aim was to demonstrate the superiority of DT pooled (20 mg/m2 and 30 mg/m2) compared to BSC treatment and not individual DT groups per protocol. OS was estimated using the Kaplan-Meier method. The comparison of treatment groups (pooled DT groups versus BSC group) was performed using a non-stratified log-rank test as the primary analysis. The Cox model and Wilcoxon test was used for sensitivity analysis; Test type: Superiority; p > 0.991, Log Rank — Treatment comparison of DT pooled with BCS used non-stratified Log-rank test at significance level p=0.05; Log rank test is used after checking the proportional hazards (PH) assumption is valid. The Wilcoxon test is used when the PH assumption fails; Hazard Ratio (HR) = 1.00 — The hazard ratio was controlled for the overall type I error rate at 5% (2-sided) corresponding to 95% confidence interval (CI) and type II error rate as 15%
Statistical Analysis 2: Comparison: Doxorubicin Transdrug (DT) 20 mg/m2 Group vs Doxorubicin Transdrug at 30 mg/m2 vs Doxorubicin Transdrug Pooled vs Best Standard of Care (BSC); Follow-up 45 month assessment: the primary aim was to demonstrate the superiority of DT pooled (20 mg/m2 and 30 mg/m2) compared to BSC treatment and not individual DT groups per protocol. OS was estimated using the Kaplan-Meier method. The comparison of treatment groups (pooled DT groups versus BSC group) was performed using a non-stratified log-rank test as the primary analysis. The Cox model and Wilcoxon test was used for sensitivity analysis; Test type: Superiority; p = 0.796, Log Rank — Treatment comparison of DT pooled with BCS used non-stratified Log-rank test at significance level p=0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.00 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from the date of randomisation to the date of the first documented progression or death from any cause. PFS determined by independent radiological review according to Response Evaluation Criteria In Solid Tumour (RECIST) 1.1 is determine by at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is considered progression.
Time Frame: Time from date of randomization to date of first documented progression or death from any cause, which ever came first, assessed up to 20 months.
Population: ITT population: All randomized patients. The DT at 20 mg/m2 and 30 mg/m2 are combined into DT pooled experimental group for comparison with the BSC group. The primary analysis is DT pooled versus BSC. This was only analyzed for the initial study.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Doxorubicin Transdrug Pooled: The DT 20 mg/m2 and 30 mg/m2 treatment group were pooled together for PFS comparison to BCS.
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Doxorubicin Transdrug Pooled | Best Standard of Care
Number analyzed (Participants) | 130 | 133 | 263 | 134
months | 2.3 [2.0 to 2.8] | 2.3 [2.1 to 2.6] | 2.3 [2.1 to 2.6] | 2.3 [2.1 to 2.8]
Statistical Analysis 1: Comparison: Doxorubicin Transdrug (DT) at 20 mg/m2 vs Doxorubicin Transdrug at 30 mg/m2 vs Best Standard of Care; PFS was estimated using Kaplan-Meier methods and plotted as curves by treatment group. For comparison between treatment groups (pooled DT 20 mg/m2 and 30 mg/m2 versus BSC) used Log-rank test as primary analysis. Hazard ratio, mean, and mean PFS rate were given with corresponding 95% CI; Test type: Superiority; p = 0.7, Log Rank — Treatment comparison with BCS using non-stratified Log-rank test at significance level p=0.05; Hazard Ratio (HR) = 1.00 — Hazard ratio for treatment variable was determined by Cox model. The hazard ratio was controlled for the overall type I error rate at 5% (2-sided) and type II error rate as 15%

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as percent of patients whose best overall response is complete response (CR) or partial response (PR) during the study treatment period and based on the evaluation of independent radiological review according to RECIST 1.1 for target lesions and assessed by MRI: CR is disappearance of all targets extra nodal lesions and the regression of all nodal lesions to < 10 mm; PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of diameters while on study. PD is at least a 20% increase in the sum of diameters of target lesions, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is considered progression.
Time Frame: Time from date of first treatment cycle to date of last cycle of treatment for the full duration of study treatment up to 24 months.
Population: ITT population: all randomized patients. The DT at 20 mg/m2 and 30 mg/m2 are combined into DT pooled experimental group for comparison with the BSC group. The primary analysis is the DT pooled versus BCS. This was only analyzed for the initial study.
Measure: Count of Participants; unit: Participants
Groups:
- Doxorubicin Transdrug at 30 mg/m2: DT will be infused over 6 hours through the IV route at dose of 30 mg/m2 on Day 1 and will be repeated every 4 weeks until disease progression or unacceptable toxicity
  Doxorubicin
- Doxorubicin Transdrug Pooled: The DT 20 mg/m2 and 30 mg/m2 treatment group were pooled together for ORR comparison to BCS.
- Best Standard of Care: Patients randomized in the control group will receive treatment according to the investigator's choice, until disease progression or unacceptable toxicity
  Best Standard of Care
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Doxorubicin Transdrug Pooled | Best Standard of Care
Number analyzed (Participants) | 130 | 133 | 263 | 134
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 2 | 2 | 1
  Stable Disease | 39 | 41 | 80 | 31
  Progressive Disease | 58 | 63 | 121 | 40
  Not Evaluable | 33 | 27 | 60 | 62
Statistical Analysis 1: Comparison: Doxorubicin Transdrug (DT) at 20 mg/m2 vs Doxorubicin Transdrug at 30 mg/m2 vs Doxorubicin Transdrug Pooled vs Best Standard of Care; The comparisons between groups (pooled DT 20 mg/m2 and 30mg/m2 versus BSC) used Fisher's exact test; Test type: Superiority; p = 1.0, Fisher Exact — Treatment comparison with BCS using Fisher's exact test at significance level p=0.05

4. Other Pre Specified Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) Considered Related to Treatment Categorized by Severity, Withdrawal From Study, or Death
Description: The number of participants experiencing TEAEs considered related to treatment and categorized by severity of all related TEAEs according to National Cancer Institute/Common Toxicity Criteria (NCI-CTCAE) v4.0 and resulting in patient withdrawal from study or death.
Time Frame: Time from date of initial treatment to date of death, disease progression, or participant withdrawal from the study.
Population: Safety Population: All patients receiving at least one infusion for DT groups and all patients for BSC group whatever treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- Best Standard of Care (BSC): Patients randomized in the control group received treatment according to the investigator's choice, until disease progression or unacceptable toxicity.
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care (BSC)
Number analyzed (Participants) | 122 | 120 | 134
Participants
  TEAEs | 79 | 98 | 58
  Severe TEAEs | 26 | 46 | 31
  Serious TEAEs | 13 | 18 | 13
  TEAEs Leading to Withdrawal | 5 | 9 | 9
  TEAEs Leading to Death | 1 | 2 | 1

5. Other Pre Specified Outcome: Number of Participants With Cardiovascular and Respiratory Events Related to Study Drug
Description: The number of participants with cardiovascular and respiratory adverse events (AEs) were assessed according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) criteria version 4.0, using the Medical Dictionary for Regulatory Activities (MedDRA). The AE numbers reported are those considered related to treatment. Related AEs are those that are judged unlikely, possibly, probably or definitely related to the study or study drug by the investigator.
Time Frame: Time from date of initial treatment to date of death, disease progression, or patient withdrawal from the study.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care (BSC)
Number analyzed (Participants) | 122 | 120 | 134
Participants
  Cardiac Disorders | 4 | 5 | 1
  Vascular Disorders | 8 | 8 | 6
  Blood Pressure Increased | 0 | 1 | 0
  Respiratory, Thoracic, and Mediastinal Disorders | 17 | 20 | 13
  Oxygen Saturation Decreased | 2 | 7 | 1
  Respiratory Rate Increased | 2 | 5 | 0
  Respiratory Rate Decreased | 1 | 1 | 0
  Ejection Fraction Decreased | 1 | 0 | 0

6. Other Pre Specified Outcome: Number of Participants Experiencing a Reduction of Oxygen Saturation (SaO2) During and After Doxorubicin Transdrug (DT) Infusion
Description: Number of participants experiencing an SaO2 reduction defined as a decrease =< 90% during or after DT infusion until resolution to =>93%. Participants had continuous monitoring of SaO2 saturation with pulse oximeter during 6 hour infusion and up to 24 hour after infusion start. SaO2 measures the amount of oxygen (in percent) bound to hemoglobin in red blood cells. SaO2 saturation was only monitored and reported in the DT infusion group. Reduction in SaO2 could result in modify DT dosing regimen. Decreases in SaO2 are a known and expected occurrence with DT infusions, and close monitoring of SaO2 was specified by the protocol to protect patients from potential respiratory distress during infusions.
Time Frame: Time from start of infusion to resolution of reduction in oxygen saturation.
Population: Safety population: All patients receiving at least one infusion for DT groups.
Measure: Count of Participants; unit: Participants
Groups:
- Doxorubicin Transdrug (DT) 20 mg/m2: DT was infused over 6 hours through the intravenous (IV) route at dose of 20 mg/m2 on Day 1 and was repeated every 4 weeks until disease progression or unacceptable toxicity.
- Doxorubicin Transdrug 30 mg/m2: DT was infused over 6 hours through the IV route at dose of 30 mg/m2 on Day 1 and was repeated every 4 weeks until disease progression or unacceptable toxicity.
Arm/Group | Doxorubicin Transdrug (DT) 20 mg/m2 | Doxorubicin Transdrug 30 mg/m2
Number analyzed (Participants) | 122 | 120
Participants | 2 | 4

7. Other Pre Specified Outcome: Number of Participants With Clinically Significant Abnormal Change in Respiratory Function
Description: Number of participants with any clinically significant abnormal change in respiratory function test over the study to include carbon monoxide diffusing capacity to measure lung function, forced expiratory volume in 1 second to measure ability to expel air from your lungs, total lung capacity to measure total amount of air in the lungs after taking the deepest breath possible, and vital capacity to measure the greatest volume of air that can be expelled from the lungs after taking the deepest breath possible. Clinically significant abnormal changes in respiratory function was determined by the investigator.
Time Frame: Time from baseline assessment to time of death, disease progression, or withdrawal of patient from the study.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care (BSC)
Number analyzed (Participants) | 122 | 120 | 134
Participants | 13 | 8 | 0

8. Other Pre Specified Outcome: Number of Participants Experiencing Clinically Significant Abnormal Electrocardiogram (ECG) Changes From Baseline
Description: Number of participants experiencing clinically significant abnormal ECG changes from baseline over the course of the study. ECG were completed every month before each infusion. ECG will detect changes in heart rhythm. Clinically significant abnormal changes in ECG were determined by the investigator.
Time Frame: Time from baseline assessment to time of death, disease progression, or withdrawal of patient from the study.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care (BSC)
Number analyzed (Participants) | 122 | 120 | 134
Participants | 4 | 6 | 5

9. Other Pre Specified Outcome: Number of Participants Experiencing Clinically Significant Changes in Left Ventricular Ejection Fraction (LVEF) and the Severity of the Event
Description: Number of participants that experienced a change from baseline in LVEF with severity of LVEF noted as follows: Normal: 100 - 50%, 0 - 9% drop from baseline resting ejection fraction (EF), Grade 2 = 50 - 40%, 10 - 19% drop from baseline resting EF; Grade 3 = 39 - 20%, >20% drop from baseline; Grade 4 = <20%. LVEF was monitored every other month. LVEF measures how much blood the left ventricle of the heart pumps out with each contraction and is used to assess the severity of left ventricle dysfunction in the heart. Clinical significance changes were determined by the investigator.
Time Frame: Time from baseline assessment to time of death, disease progression, or withdrawal of patient from the study.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care (BSC)
Number analyzed (Participants) | 122 | 120 | 134
Participants
  At Least One Abnormal Value | 1 | 4 | 2
  At Least One Grade 3-4 Value | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected until 1 month after last treatment. Treatment continued until patient experienced disease progression, aggravation of liver dysfunction, death, serious AE (SAE), or intolerable AE; or the patient withdrew consent or was withdrawn from study by investigator for reasons listed in the protocol. Median treatment durations were 1.9, 2.7, and 2.4 months in the Doxorubicin Transdrug (DT) 20 mg/m2, DT 30 mg/m2, and best standard of care (BSC) groups, respectively.
Description: The incidence and severity of all AEs and SAEs were assessed according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) criteria version 4.0, using the Medical Dictionary for Regulatory Activities (MedDRA). The cutoff for AE reporting was May 28, 2017.
Arm/Group | Doxorubicin Transdrug (DT) at 20 mg/m2 | Doxorubicin Transdrug at 30 mg/m2 | Best Standard of Care
All-Cause Mortality (participants affected / at risk) | 118/122 | 119/120 | 113/134
Serious Adverse Events (participants affected / at risk) | 37/122 | 37/120 | 48/134
Other Adverse Events (participants affected / at risk) | 110/122 | 112/120 | 97/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin Transdrug (DT) at 20 mg/m2 (N=122) | Doxorubicin Transdrug at 30 mg/m2 (N=120) | Best Standard of Care (N=134)
Catheter site infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 2 (2) | 8 (8)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 5 (6) | 7 (9)
Oxygen saturation decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Respiratory rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 7 (7)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Complications associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Coma hepatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Venous ulcer pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired quality of life (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin Transdrug (DT) at 20 mg/m2 (N=122) | Doxorubicin Transdrug at 30 mg/m2 (N=120) | Best Standard of Care (N=134)
Asthenia (General disorders) | 41 (65) | 57 (82) | 39 (48)
Fatigue (General disorders) | 9 (11) | 14 (18) | 14 (15)
Pyrexia (General disorders) | 9 (13) | 23 (32) | 8 (8)
Nausea (Gastrointestinal disorders) | 26 (44) | 33 (62) | 24 (28)
Diarrhoea (Gastrointestinal disorders) | 21 (39) | 23 (31) | 20 (26)
Vomiting (Gastrointestinal disorders) | 15 (19) | 20 (28) | 10 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 14 (26) | 24 (40)
Anaemia (Blood and lymphatic system disorders) | 15 (24) | 22 (30) | 22 (28)
Neutropenia (Blood and lymphatic system disorders) | 4 (16) | 18 (41) | 7 (9)
Leukopenia (Blood and lymphatic system disorders) | 1 (6) | 11 (23) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 5 (6) | 7 (16) | 3 (4)
Paraesthesia (Nervous system disorders) | 4 (5) | 2 (2) | 20 (35)
Headache (Nervous system disorders) | 11 (12) | 16 (23) | 6 (8)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 9 (9)
Decreased Appetite (Metabolism and nutrition disorders) | 16 (16) | 19 (19) | 21 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 7 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (20) | 12 (16) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 9 (10) | 10 (12)
Oedema peripheral (General disorders) | 9 (10) | 25 (27) | 24 (26)
Mucosal inflammation (General disorders) | 2 (2) | 6 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 18 (22) | 15 (18) | 12 (14)
Abdominal pain (Gastrointestinal disorders) | 13 (15) | 15 (18) | 13 (17)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 12 (15) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 11 (13) | 5 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (9) | 6 (13) | 6 (11)
Weight decreased (Investigations) | 5 (5) | 13 (13) | 5 (5)
Blood bilirubin increased (Investigations) | 8 (9) | 2 (3) | 7 (12)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 6 (6) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10) | 9 (10) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 3 (3)
Dizziness (Nervous system disorders) | 7 (8) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 15 (23) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) | 5 (5)
Bronchitis (Infections and infestations) | 7 (10) | 7 (7) | 4 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 7 (17) | 3 (3)
Jaundice (Hepatobiliary disorders) | 2 (2) | 8 (9) | 1 (1)
Hypertension (Vascular disorders) | 8 (10) | 5 (5) | 3 (5)
Anxiety (Psychiatric disorders) | 3 (3) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT01655693/Prot_SAP_000.pdf